CLINICAL TRIAL: NCT05493917
Title: A Real-world Study to Evaluate the Safety and Immunogenicity of a Third-dose Booster After Two Doses of an Inactivated COVID-19 Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, chief physician, Huashan Hospital
Other Study IDs: KY2021-923
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Vaccine Reaction
Keywords: inactive vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: an inactivated SARS-CoV-2 vaccine named BBIBP-CorV — Completed 2 doses of an inactivated SARS-CoV-2 vaccine more than 6 months ago and received a third dose of the vaccine

SUMMARY:
This project is a prospective observational real-world study, recruiting and screening subjects who have completed 2 doses of the COVID-19 vaccine for more than 6 months and receive the third dose of the vaccine voluntarily into the clinical cohort of this study. Subjects received a third dose of the COVID-19 vaccine will be enrolled in the study and followed up for 1 year at baseline (day 0) before vaccine injection, 28 days after injection, 90 days, 270 days after injection. On the 365th day, blood samples were collected for the detection of anti-SARS-CoV-2 antibodies and other related indicators to evaluate the immune protection effect.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old, gender is not limited;
* Subjects who completed the second dose of COVID-19 inactivated vaccine for more than 6 months and received the third dose of the same vaccine

Exclusion Criteria:

* allergic to the active ingredients of the SARS-CoV-2 vaccine, any of the inactive ingredients, the substances used in the production process, or those who have had allergies during previous vaccination of similar vaccines;
* those who have had severe allergic reactions to vaccines in the past (such as acute allergic reactions, angioedema, respiratory Difficulties, urticaria, angioedema or abdominal pain);
* Receiving other research drugs within 3 months ;participating in other research vaccines Or subjects in clinical trials of research drugs;
* other conditions that the investigator judges are not suitable for this clinical trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruit and screen subjects who have completed 2 doses of the new coronavirus vaccine for more than 6 months and voluntarily receive a third dose of the vaccine
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) | Day 28±3 after the third dose of vaccine injection
  Geometric mean titers (GMTs) of serum COVID-19 neutralizing antibodies

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) | Day 90±7, Day 180±7, Day 270±7, Day 365±7 after the third dose of vaccine injection
  Geometric mean titers (GMTs) of serum COVID-19 neutralizing antibodies
IgG | Day 28±3, Day 90±7, Day 180±7, Day 270±7, Day 365±7 after the third dose of vaccine injection
  Serum SAS-CoV-2 IgG

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious department of Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No